CLINICAL TRIAL: NCT04311463
Title: An Oral Single-dose, Randomized, Balanced, Open-label, Two-sequence, Two-treatment, Two-period, Crossover Bioequivalence Study of Paroxetine Tablets 20 mg of GlaxoSmithKline Pharmaceuticals S.A, With That of PAXIL (Paroxetine) Tablets 20 mg of GlaxoSmithKline México S.A. de C.V., in Healthy Adult Male and Female Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Paroxetine and PAXIL Under Fasting Conditions in Healthy Mexican Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 212969
Record Dates: First submitted 2020-03-16; First posted 2020-03-17 (Actual); Results first posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-12

CONDITIONS: Anxiety Disorders
Keywords: Anxiety Disorders; Bioequivalence study; Paroxetine hydrochloride; PAXIL; Fasting condition
MeSH Terms: conditions — Anxiety Disorders | interventions — Paroxetine

STUDY DESIGN:
Intervention Model Description: A single-dose, randomized, balanced, open-label, two-sequence, two-treatment, two-period, crossover bioequivalence study under fasting condition.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paroxetine hydrochloride followed by PAXIL (Experimental)
  Interventions: Drug: Paroxetine hydrochloride; Drug: PAXIL (Paroxetine hydrochloride )
- PAXIL followed by paroxetine hydrochloride (Experimental)
  Interventions: Drug: Paroxetine hydrochloride; Drug: PAXIL (Paroxetine hydrochloride )

INTERVENTIONS:
Drug: Paroxetine hydrochloride — Paroxetine hydrochloride will be administered.
Drug: PAXIL (Paroxetine hydrochloride ) — PAXIL will be administered.

SUMMARY:
This study will be conducted to evaluate and compare the single oral dose bioavailability of Paroxetine manufactured by GlaxoSmithKline (GSK) Pharmaceuticals S.A. for GlaxoSmithKline México, S.A. de C.V. with that of PAXIL® (Paroxetine) of GlaxoSmithKline, México, S.A. de C.V. in healthy, adult, male and female participants under fasting conditions. Maximum 38 participants will be randomized and dosed. The expected duration of this study will be 12 days including 7 days of washout period in-between each dosing. PAXIL is a registered trademark of GSK group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female participants aged between 18 and 55 years.
* Participant is a light smoker (someone who smokes 9 or less cigarettes per day) or non- or an ex-smoker (someone who completely stopped smoking for at least 6 months before day 1 of this study).
* With a weight greater than or equal to (>=)50.00 kilograms (kg).
* With a body mass index (BMI) >=18.5 kilograms per meter square (kg/m^2) and less than or equal to (<=)27.0 kg/m^2.
* Found healthy according to the clinical laboratory results and physical examination (performed within 90 days prior to the dosing on period -1).
* Have a normal 12 lead electrocardiogram (ECG) and vital signs.
* Have laboratory test results within the laboratory's stated normal range; if not within this range, they must lack of no clinical significance as judged by the principal investigator (PI) or responsible physician.
* Willing to avoid sexual contact or use an acceptable contraceptive method during the study including the washout period (for females). In case of male participants, they should avoid sexual contact or use a latex or synthetic condom each time they have sex with a woman while taking Paroxetine and during 7 days after the end of the study.
* If study participant is a female and is of child bearing potential, practicing an acceptable method of birth control for the duration of the study as judged by the investigators, like combined short acting (estrogen and progestogen containing) hormonal contraception for example (e.g.) oral, intravaginal, and progestogen-only hormonal contraception e.g. oral, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), condoms, foams, jellies and diaphragm or abstinence or if study participant is a female and is postmenopausal for at-least 1 year or is surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has been performed on the study participant).
* Have a negative test for active Coronavirus Disease-2019 (COVID-19), within 72 hours prior to the first period check-in. The testing should be done using a molecular (Real time-Polymerase Chain Reaction [RT-PCR]) approved by the country regulatory authorities.
* Participant is able to communicate effectively and voluntarily agreed to participate in this study by signing written informed consent after being informed sufficiently about study aspects like objectives, study procedures, characteristics of the investigational drug, expected adverse events.
* Participant willing to adhere to protocol requirements as described in informed consent (written) approved by research ethics committee/research committee (REC/RC).

Exclusion Criteria:

* If participants age is less than 18 or older than 55 years.
* Have any history of allergy or hypersensitivity to Paroxetine or derivatives to any of its metabolites/derivatives or related drugs or excipients.
* Have a positive test result for hepatitis B surface antigen (HBs Ag) or hepatitis C virus antibody (HCV Ab) or human immune deficiency virus (HIV) antibodies (types 1 and 2) or venereal disease research laboratory (VDRL).
* Participants with symptoms suggestive of active COVID-19 infection (that is, fever, cough, respiratory difficulties) within 14 days of inpatient admission.
* Participants with known COVID-19 positive contact (meaning if the participant has been living, providing care, being within 1.5 meters for at least 15 min or having exposure to respiratory secretions with/to a person who has COVID-19) within the past 14 days prior to the first period check-in. Study drug is contraindicated for medical reasons to the participants.
* Have any history or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, seizures, endocrine, dermatological, neurological or psychiatric disease or disorder (e.g. participants with uncontrolled hypertension, pheochromocytoma, carcinoid, thyrotoxicosis, bipolar depression, schizoaffective disorder and acute confusional states).
* Presence of significant gastrointestinal, hepatic or kidney disease, or surgery or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects or participants with a history of gastrointestinal disorder or surgery which may affect the absorption of investigational drug.
* Have a history of alcohol abuse or drug abuse during the last 1 year prior to period -1 dosing.
* Have a history of smoking >=10 cigarettes per day during the last 6 months prior to period -1 dosing.
* Have history or presence of cancer.
* Have any history of gastrointestinal ulcers/intestinal bleeding.
* Have history of difficulty for donating blood.
* Have clinically significant abnormal laboratory tests results.
* Have a systolic blood pressure less than (<)90 or greater than (>)140 millimeters of mercury (mmHg) or diastolic blood pressure is <60 or >90 mmHg.
* Have a pulse rate <60 beats/minute or >100 beats/minute (lower range of pulse range will be accepted up to 45 beats/minute in case of athlete).
* Have used any prescribed medication during the last 14 days preceding the first dosing, or use over-the-counter (OTC), medicinal or herbal products during the last 7 days or use medicinal enzyme inhibitors / inducers during last 30 days preceding the first dosing.
* Have participated in a drug research study or donated blood within the last 3 months.
* Have a positive result for drugs of abuse test (cannabinoids [marijuana/tetrahydrocannabinol-(THC)], cocaine, opiates/morphine, amphetamine, methamphetamine and benzodiazepines] performed during screening.
* Female participant, who is currently breast feeding or a who is pregnant or who is likely to become pregnant during the study.
* Female participant has a positive pregnancy test results.
* Unwillingness or inability to comply with the instructions on the lifestyle.
* If the PI considers, for any reason, that the volunteer is not a suitable candidate to receive the study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-dose, randomized, balanced, open-label, two-sequence, two-treatment, two-period, crossover bioequivalence study of Paroxetine tablets 20 milligrams (mg) of GlaxoSmithKline (GSK) Pharmaceuticals S.A, with that of PAXIL (Paroxetine) tablets 20 mg of GSK México S.A. de C.V., in healthy adult male & female participants under fasting conditions.
Pre-assignment Details: Total 38 participants were enrolled in the study across one study center in Mexico.
Groups:
- Paroxetine 20 mg (A) Followed by Paxil 20 mg (B): Participants received Paroxetine 20 mg tablet (Test drug A) as a single oral dose in treatment period 1. In treatment period 2, participants received Paxil 20 mg tablet (Reference drug B) as a single oral dose. There was a washout period of atleast 7 days between two treatment periods.
- Paxil 20 mg (B) Followed by Paroxetine 20 mg (A): Participants received Paxil 20 mg tablet (Reference drug B) as a single oral dose in treatment period 1. In treatment period 2, participants received Paroxetine 20 mg tablet (Test drug A) as a single oral dose. There was a washout period of atleast 7 days between two treatment periods.
Period: Period 1 (Up to Day 3)
Arm/Group | Paroxetine 20 mg (A) Followed by Paxil 20 mg (B) | Paxil 20 mg (B) Followed by Paroxetine 20 mg (A)
Started | 19 | 19
Completed | 18 | 19
Not Completed | 1 | 0
Not completed — Participant met Protocol defined withdrawal criteria | 1 | 0
Period: Washout Period (Up to Day 7)
Arm/Group | Paroxetine 20 mg (A) Followed by Paxil 20 mg (B) | Paxil 20 mg (B) Followed by Paroxetine 20 mg (A)
Started | 18 | 19
Completed | 17 | 18
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Period 2 (Up to Day 3)
Arm/Group | Paroxetine 20 mg (A) Followed by Paxil 20 mg (B) | Paxil 20 mg (B) Followed by Paroxetine 20 mg (A)
Started | 17 | 18
Completed | 15 | 17
Not Completed | 2 | 1
Not completed — Participant met Protocol defined withdrawal criteria | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine 20 mg (A) Followed by Paxil 20 mg (B) | Paxil 20 mg (B) Followed by Paroxetine 20 mg (A) | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 10 | 13 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Paroxetine
Description: Blood samples were collected at indicated time points for the analysis of Cmax of Paroxetine. PK parameters were analyzed using non-compartmental analysis.
Time Frame: Pre-dose (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 9, 10, 12, 16, 24, 36, 48 and 72 hours post-dose
Population: Pharmacokinetic (PK) analysis set included participants who completed both period of the study as per protocol criteria. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Groups:
- Paroxetine 20 mg (Test A): Participants received Paroxetine 20 mg (Test A) as a single oral dose in fasting condition in Periods 1 and 2
- Paroxetine 20 mg (Reference B): Participants received Paxil (Paroxetine) 20 mg (Reference B) as a single oral dose in fasting condition in Periods 1 and 2.
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
Number analyzed (Participants) | 31 | 31
Nanograms per milliliter | 8.39 (5.872) | 8.83 (6.554)

2. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to the Last Measurable Concentration (AUC[0-t]) of Paroxetine
Description: Blood samples were collected at indicated time points for the analysis of AUC(0-t) of Paroxetine. PK parameters were analyzed using non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Hour*nanograms per milliliter
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
Number analyzed (Participants) | 31 | 30
Hour*nanograms per milliliter | 128.876 (118.288) | 150.549 (137.497)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of Paroxetine
Description: Blood samples were collected at indicated time points for the analysis of AUC(0-inf) of Paroxetine. PK parameters were analyzed using non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Hour*nanograms per milliliter
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
Number analyzed (Participants) | 31 | 30
Hour*nanograms per milliliter | 142.482 (149.098) | 160.143 (149.403)

4. Primary Outcome: Percentage of AUC (0 to Infinity) Obtained by Extrapolation (%AUCex) of Paroxetine
Description: Blood samples were collected at indicated time points for the analysis of %AUCex of Paroxetine. PK parameters were analyzed using non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of AUCex
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
Number analyzed (Participants) | 31 | 30
Percentage of AUCex | 7.95 (8.053) | 7.05 (7.499)

5. Primary Outcome: Time of the Maximum Measured Plasma Concentration (Tmax) of Paroxetine
Description: Blood samples were collected at indicated time points for the analysis of Tmax of Paroxetine. PK parameters were analyzed using non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
Number analyzed (Participants) | 31 | 31
Hours | 5.00 [1.50 to 8.00] | 5.00 [0 to 8.00]

6. Primary Outcome: Elimination Half-life (t1/2) of Paroxetine
Description: Blood samples were collected at indicated time points for the analysis of t1/2 of Paroxetine. PK parameters were analyzed using non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
Number analyzed (Participants) | 31 | 30
Hours | 10.78 [4.19 to 21.46] | 11.32 [7.96 to 21.32]

7. Primary Outcome: Terminal Elimination Rate Constant (Kel) of Paroxetine
Description: Blood samples were collected at indicated time points for the analysis of Kel of Paroxetine. PK parameters were analyzed using non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Per hour
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
Number analyzed (Participants) | 31 | 30
Per hour | 0.0653 (0.02152) | 0.0618 (0.01331)

8. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence that may occur in a research participant during clinical research phase of a drug or vaccine but which does not necessarily has a causal relationship with this. SAE is defined as any medical occurrence that, at any dose, put participants's life in risk or results in death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent significant disability/incapacity, is a congenital anomaly/birth defect and other important medical events according to medical or scientific judgement.
Time Frame: Up to 25 days
Population: Safety analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
Number analyzed (Participants) | 38 | 38
Participants
  Non-serious AEs | 7 | 7
  SAEs | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse rate, respiration rate and body temperature were measured in semi-supine position after 5 minutes rest. The clinically acceptable range included; SBP: 85 millimeters of mercury (mmHg) to 160 mmHg; DBP: 45 mmHg to 100 mmHg; pulse rate: 40 beats per minute to 110 beats per minute; respiration rate: 8 breaths per minute to 20 breaths per minute; body temperature: 35.5 degrees Celsius to 37.8 degrees Celsius. Number of participants with any abnormality in vital signs are presented. Data is presented treatment wise.
Time Frame: Up to 25 days
Population: Safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
Number analyzed (Participants) | 38 | 38
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious AEs and Serious AEs were collected up to 25 days
Description: All-cause mortality, non-serious AEs and SAEs were collected in safety analysis set. Safety analysis set included all participants who received at least one dose of study treatment.
Arm/Group | Paroxetine 20 mg (Test A) | Paroxetine 20 mg (Reference B)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 7/38 | 7/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine 20 mg (Test A) (N=38) | Paroxetine 20 mg (Reference B) (N=38)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Nervous system disorders) | 3 (3) | 4 (5)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 5 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT04311463/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT04311463/SAP_001.pdf